CLINICAL TRIAL: NCT00227240
Title: Observational Study With Enbrel (Etanercept) in Adult Patients With Plaque Psoriasis
Brief Title: Study Evaluating Enbrel (Etanercept) in Adult Patients With Plaque Psoriasis
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A-101789
Record Dates: First submitted 2005-09-13; First posted 2005-09-27 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to investigate the incidences of adverse events for patients with plaque psoriasis treated with Enbrel under usual care settings.

ELIGIBILITY:
Inclusion Criteria:

* Proven diagnosis of Plaque Psoriasis

Exclusion Criteria:

* Contraindications according to SmPC of Enbrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinical and community sample
Sampling Method: Non-Probability Sample
Enrollment: 753 (Actual)
Dates: Start 2005-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Germany (2):
  - Pfizer Investigational Site, Munich
  - Pfizer Investigational Site, München

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A-101789&StudyName=Study%20Evaluating%20Enbrel%20%28Etanercept%29%20in%20adult%20patients%20with%20plaque%20psoriasis